CLINICAL TRIAL: NCT01604252
Title: A Prospective Observational Study of Treatment Patterns and Effectiveness and Safety Outcomes in Advanced Basal Cell Carcinoma and Basal Cell Carcinoma Nevus Syndrome Patients
Brief Title: An Observational Study of Treatment Patterns and Effectiveness and Safety Outcomes in Advanced Basal Cell Carcinoma and Basal Cell Carcinoma Nevus Syndrome Patients(RegiSONIC)
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early by the Sponsor due to the high rate of discontinuation of subjects unrelated to patient safety.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28296
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — optional blood sample

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, prospective, observational cohort study will evaluate the effectiveness, safety and utilization of treatments in patients with advanced basal cell carcinoma and basal cell carcinoma nevus syndrome. The total study duration is anticipated to be a maximum of 8 years, including 3 years for patient recruitment and 5 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with basal cell carcinoma (BCC) who meet either of the following definitions:

  * Patients who were determined with advanced disease (aBCC) within 90 days prior to study enrollment, have not been diagnosed with basal cell carcinoma nevus syndrome (BCCNS) and have not been treated with an investigational or approved hedgehog pathway inhibitor
  * Patients with aBCC who have not been diagnosed with BCCNS and who were previously treated with vismodegib as part of Genentech study SHH4476g, SHH4437g, or SHH4811g (EAP)
  * Patients with BCCNS who either have aBCC or multiple BCCs of any stage as defined by protocol (may include patients previously enrolled in Genentech study SHH4476g, SHH4437g, or SHH4811g (EAP))

Exclusion Criteria:

* Participation in a clinical trial within 90 days prior to study enrollment that has either involved treatment of aBCC or involved treatment with an investigational or approved hedgehog pathway inhibitor, except for patients treated with vismodegib as part of Genentech study SHH4476g, SHH4437g, or SHH4811g (EAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for advanced basal cell carcinoma and basal cell carcinoma nevus syndrome
Sampling Method: Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Response rate | approximately 5 years
Duration of response | approximately 5 years
Recurrence rate | approximately 5 years
Progression-free survival | approximately 5 years
Overall survival | approximately 5 years
Safety: Incidence of adverse events | approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (81):
- United States (80):
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Moy-Fincher-Chipps Facial Plastics and Dermatology, Beverly Hills, California
  - University of California Irvine, Irvine, California
  - Scripps Clinic; Hematology & Oncology, La Jolla, California
  - University of California San Diego, La Jolla, California
  - Fairmont Dermatology Medical Associates, Inc., Lodi, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Dermatology Research Associate, Los Angeles, California
  - Newport Dermatology and Laser Associates, Newport Beach, California
  - Stanford University, Palo Alto, California
  - Skin Surgery Med Group, Inc, San Diego, California
  - University Clinical Trials, San Diego, California
  - Clinical Research Specialists, Inc., Santa Monica, California
  - California Pacific Medical Center Research Institute, Santa Rosa, California
  - Pacific Dermatology Institute, Temecula, California
  - Advanced Derm & Cosmetic Care, Valencia, California
  - University of Colorado; Anschutz Cancer Pavilion, Aurora, Colorado
  - Dermatology Associates and Research, Coral Gables, Florida
  - NOVA Southeastern University, Fort Lauderdale, Florida
  - Hollywood Dermatology and Cosmetic Specialists, Hollywood, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Advanced Derm & Cosmetic Surg, Ormond Beach, Florida
  - Belleair Research Center, Pinellas Park, Florida
  - Skin and Cancer Associates and the Center for Cosmetic Enhancement, Plantation, Florida
  - Florida Research Specialists, Seminole, Florida
  - Spencer Derma & Skin Surg Ctr, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Inst., Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Kenneth R. Beer, M.D., PA, West Palm Beach, Florida
  - Georgia Skin Cancer and Aesthetic Dermatology, Athens, Georgia
  - Emory Univ Winship Cancer Inst, Atlanta, Georgia
  - Dermatologic Surgery Specialists, Inc, Macon, Georgia
  - Northwest Georgia Dermatology and Skin Cancer Specialists, Marietta, Georgia
  - Gwinnett Clinical Research Center, Snellville, Georgia
  - Northwestern University, Chicago, Illinois
  - Southern IL Univ School of Med, Springfield, Illinois
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Shideler Clinical Research Center, Carmel, Indiana
  - Indiana Clinical Trial Center, Plainfield, Indiana
  - MLF Knuckles, MD, PSC, Corbin, Kentucky
  - Derm Research, LLC, Louisville, Kentucky
  - Beverly Hospital, A Member of Lahey Health, Beverly, Massachusetts
  - Faulkner Hospital, Jamaica Plain, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota., Minneapolis, Minnesota
  - University of Mississippi Medical Center; Division of Dermatology, Jackson, Mississippi
  - Laser and Dermatologic Surgery Center, Chesterfield, Missouri
  - Saint Louis University School of Medicine; Department of Dermatology, St Louis, Missouri
  - Associated Dermatology and Skin Cancer Clinic of Helena, PC, Helena, Montana
  - Bettencourt Skin Center, Henderson, Nevada
  - Linda Woodson Dermatology, A Professional Corporation, Las Vegas, Nevada
  - Woodson Dermatology, Las Vegas, Nevada
  - Strimling Dermatology, Laser and Vein Institute, Las Vegas, Nevada
  - Skin Cancer and Dermatology Institute, Reno, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Dermatology Group, P.C., Verona, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Long Island Skin Cancer and Dermatologic Surgery, Smithtown, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Skin Surgery Center, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University; Comp Can Ctr, Columbus, Ohio
  - University of Oklahoma Health Sciences Cente; Department of Dermatology, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Dermatology and Laser Center of Charleston PA, Charleston, South Carolina
  - The Sarah Cannon Research Inst, Nashville, Tennessee
  - DermSurgery Associates, PA, Houston, Texas
  - South Texas Research Alliance LLC, Laredo, Texas
  - South Valley Dermatology Center, West Jordan, Utah
  - Dermatology Associates PLLC, Seattle, Washington
  - Huntington Internal Medicine Group, Huntington, West Virginia
  - Manish J. Gharia, MD, Brookfield, Wisconsin
- Alma M Cruz MD, Carolina, Puerto Rico